CLINICAL TRIAL: NCT06594627
Title: Smart Pillows for Enhancing Sleep Quality_Pilot Study
Brief Title: Smart Pillows for Enhancing Sleep Quality
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Chang Dae Lee, Assistant Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22402
Record Dates: First submitted 2024-09-03; First posted 2024-09-19 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Snoring; Obstructive Sleep Apnea
Keywords: assistive device; sleep quality; snoring; obstructive sleep apnea
MeSH Terms: conditions — Snoring; Sleep Apnea, Obstructive; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: It is a single group, pre- and post- test/eval design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Smart pillow group (Experimental): There is one group that will receive an intervention: the utilization of a smart pillow to mitigate snoring issues and OSA symptoms.
  Interventions: Device: Smart pillow

INTERVENTIONS:
Device: Smart pillow — Utilize a smart pillow that is designed to reduce snoring issues and OSA symptoms during sleep
  Other Names: Nitetronic Z6 smart pillow

SUMMARY:
The purpose of this study is to examine the impact of smart pillows on the sleep quality of individuals who experience a snoring issue and/or obstructive sleep apnea (OSA), as well as their sleep partners. Furthermore, this study will explore whether enhancements in sleep quality positively influence depressive symptoms, physical activity, heart rate, blood oxygen levels, and cognitive functions.

DETAILED DESCRIPTION:
The study's timeline consists of 3 phases:

* a pre-evaluation, or baseline, phase during the 7 days prior to study pillow use,
* an intervention phase, occurring for 14 days during study pillow use,
* a post-evaluation phase, during the final 7 days of study pillow use.

During the Pre-Evaluation phase, participants and their sleep partners will complete questionnaires related to sleep quality and depression. Participants and sleep partners will each be asked to wear an actigraphy watch continuously for the 7 days immediately prior to the intervention phase (Study Day -7 through Study Day -1). The actigraphy watch will collect data on various objective sleep quality measures and on other health measures. Additionally, participants and sleep partners will also complete a daily sleep log and a daily sleep questionnaire during this pre-evaluation phase. The participant (individual with snoring or OSA) will also set up the pillow's control box next to the bed to collect baseline data on snoring patterns.

During the Intervention phase, participants with snoring issues or OSA will be asked to use the study pillow for 14 days (Study Day 1 through Study Day 14). The pillow features a center that detects the head position and six airbags that can add and remove air individually. If the pillow detects snoring, it will adjust the position of the participant's head by adjusting the amount of air in each airbag. This repositioning is gentle, produces minimal noise, and will not disrupt the participant's sleep or wake them. Participants will be provided with instructions on how to use the pillow. Participants may continue current snoring or OSA treatments during this time. During the intervention phase, sleep partners will be asked to continue to share a sleeping space with the participant, as they are used to doing.

The post-evaluation phase begins half-way through the intervention phase and continues through discontinuation of the study pillow (Study Day 8 through Study Day 14). During the post-evaluation phase, participants and sleep partners will repeat the assessments from the Pre-Evaluation phase, including the daily wear of the actigraphy watch and the daily sleep log and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for individuals with snoring issues or OSA

  * Individuals 50 years of age or older.
  * Individuals who experience snoring issues and/or OSA that may impact their perceived sleep quality or that of their sleep partner.
  * Individuals who currently use and do not use snoring and/or OSA treatment (participants will not be asked or required to discontinue any current snoring and/or OSA treatments that they are prescribed or using.)
  * Individuals who have a smartphone or a smart mobile device (Apple iOS 15 and higher or Android 10 or higher).
  * Individuals with and without a sleep partner.
  * Individuals who do not have a pacemaker.
  * Individuals who do not have intracranial electrodes.
  * Individuals who do not have neck pain related to the cervical spine problems, including disc, muscle, and neurological issues.

Inclusion criteria for sleep partners

* Individuals aged 18 years and older.
* Individuals who share the same sleeping space with their sleep partner (who has snoring issues and/or OSA) more than four times a week.
* Individuals whose sleep partner (who has snoring issues and/or OSA) agrees to participate in this study.

Exclusion Criteria:

* Any participant who is not able to consent or complete study interventions independently, as determined by the investigator.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-11-18 (Actual); Primary Completion 2026-07-11 (Estimated); Study Completion 2026-07-11 (Estimated)

PRIMARY OUTCOMES:
Change in Participant Subjective Sleep Quality (PSQI) | Baseline and Day 14
  Subjective sleep quality will be measured by the Pittsburgh Sleep Quality Index (PSQI). The PSQI score ranges from 0-21. A higher score indicates worse sleep quality. The PSQI will be administered prior to use of the study pillow and again after discontinuing use of the study pillow.
Change in Participant Subjective Sleep Quality (novel sleep quality questionnaire) | Day -7 through Day -1 and Day 8 through Day 14
  Subjective sleep quality will also be measured by a novel questionnaire created for this project. Questionnaire score ranges from 3-15. A higher score indicates better sleep quality. Participants will be asked to complete this questionnaire 14 times during their participation: once daily for the 7 days prior to initiating use of the study pillow (Day -7 through Day -1) and once daily for the last 7 days of study pillow use (Day 8 - Day 14).
Change in Participant total sleep time | Day -7 through Day -1 and Day 8 through Day 14
  As part of measuring objective sleep quality, total sleep time will be measured using the Fitbit Inspire 3 (an actigraphy watch). Participants will be asked to wear the actigraphy watch continuously for the 7 days before initiating use of the study pillow (Day -7 through Day -1) and continuously for the last 7 days of study pillow use (Day 8 through Day 14).
Change in Participant sleep periods | Day -7 through Day -1 and Day 8 through Day 14
  As part of measuring objective sleep quality, sleep periods (light and deep sleep) will be measured using the Fitbit Inspire 3 (an actigraphy watch). Participants will be asked to wear the actigraphy watch continuously for the 7 days before initiating use of the study pillow (Day -7 through Day -1) and continuously for the last 7 days of study pillow use (Day 8 through Day 14).
Change in Participant REM sleep time | Day -7 through Day -1 and Day 8 through Day 14
  As part of measuring objective sleep quality, REM and non-REM sleep time will be measured using the Fitbit Inspire 3 (an actigraphy watch). Participants will be asked to wear the actigraphy watch continuously for the 7 days before initiating use of the study pillow (Day -7 through Day -1) and continuously for the last 7 days of study pillow use (Day 8 through Day 14).
Change in Participant Snoring time | Days 1 - 14 (during use of the study pillow)
  The study pillow (Nitetronic Z6 smart pillow) will collect data on total time spent snoring and the intensity of the snoring. Participants will be asked to use the study pillow for 14 consecutive nights during their participation (Day 1 through Day 14).
Change in Participant Depressive symptoms | Baseline and Day 14
  Depressive symptoms will be measured using the Center for Epidemiologic Studies Depression Scale, 8-item (CES-D-8). The CES-D-8 score ranges from 0 to 8. A higher score indicates more severe depressive symptoms.. The CES-D-8 will be administered prior to use of the study pillow and again after discontinuing use of the study pillow.
Change in Participant blood oxygen level | Day -7 through Day -1 and Day 8 through Day 14
  Blood oxygen level will be measured using the Fitbit Inspire 3 (an actigraphy watch). Participants will be asked to wear the actigraphy watch continuously for the 7 days before initiating use of the study pillow (Day -7 through Day -1) and continuously for the last 7 days of study pillow use (Day 8 through Day 14).
Change in Participant physical activity level | Day -7 through Day -1 and Day 8 through Day 14
  Physical activity level will be measured using the Fitbit Inspire 3 (an actigraphy watch). Participants will be asked to wear the actigraphy watch continuously for the 7 days before initiating use of the study pillow (Day -7 through Day -1) and continuously for the last 7 days of study pillow use (Day 8 through Day 14).
Change in Participant's subjective cognitive function | Baseline and Day 14
  Subjective cognitive function will be measured by a two-question questionnaire: 1) 'How would you rate your memory at the present time? Would you say it is excellent, very good, good, fair, or poor?' and 2) 'Compared to the previous month, would you say your memory is better now, about the same, or worse than it was then?' The two-question questionnaire will be administered prior to the use of the study pillow and again after discontinuing the use of the study pillow.
Change in Participant's objective cognitive function | Baseline and Day 14
  Objective cognitive function will measured by the Montreal Cognitive Assessment (MoCA). The MoCA score ranges from 0-30. A higher score indicates better cognitive function. The MoCA will be administered prior to the use of the study pillow and again after discontinuing the use of the study pillow.

SECONDARY OUTCOMES:
Change in Partner's Subjective Sleep Quality (PSQI) | Baseline and Day 14
  Subjective sleep quality will be measured by the Pittsburgh Sleep Quality Index (PSQI). The PSQI score ranges from 0-21. A higher score indicates worse sleep quality. The PSQI will be administered to sleep partners of study participants prior to the participant's use of the study pillow and again after the participant discontinues use of the study pillow.
Change in Partner's Subjective Sleep Quality (novel sleep quality questionnaire) | Days -7 through -1 and Days 8-14
  Subjective sleep quality will also be measured by a novel questionnaire created for this project. Questionnaire score ranges from 3-15. A higher score indicates better sleep quality. Sleep Partners will be asked to complete this questionnaire 14 times during their participation: once daily for the 7 days prior to the participant initiating use of the study pillow (Day -7 through Day -1) and once daily during the participant's last 7 days of study pillow use (Day 8 through Day 14).
Change in Partner's total sleep time | Day -7 through Day -1 and Day 8 through Day 14
  As part of measuring objective sleep quality, total sleep time will be measured using the Fitbit Inspire 3 (an actigraphy watch). Sleep Partners of study participants will be asked to wear the actigraphy watch continuously for 7 days before the participant initiates use of the pillow (Day -7 through Day -1) and continuously for the last 7 days of the participant's pillow use (Day 8 through Day 14).
Change in Partner's sleep periods | Day -7 through Day -1 and Day 8 through Day 14
  As part of measuring objective sleep quality, sleep periods (light and deep sleep) will be measured using the Fitbit Inspire 3 (an actigraphy watch). Sleep Partners of study participants will be asked to wear the actigraphy watch continuously for the 7 days before the participant initiates use of the pillow (Day -7 through Day -1) and continuously for the last 7 days of the participant's pillow use (Day 8 through Day 14).
Change in Partner's REM sleep time | Day -7 through Day -1 and Day 8 through Day 14
  As part of measuring objective sleep quality, REM and non-REM sleep time will be measured using the Fitbit Inspire 3 (an actigraphy watch). Sleep Partners of study participants will be asked to wear the actigraphy watch continuously for the 7 days before the participant initiates use of the pillow (Day -7 through Day -1) and continuously for the last 7 days of the participant's pillow use (Day 8 through Day 14).
Change in Partner Depressive symptoms | Baseline and Day 14
  Depressive symptoms will be measured using the Center for Epidemiologic Studies Depression Scale, 8-item (CES-D-8). The CES-D-8 score ranges from 0 to 8. A higher score indicates more severe depressive symptoms. The CES-D-8 will be administered prior to use of the study pillow and again after discontinuing use of the study pillow.
Change in Partner's blood oxygen level | Day -7 through Day -1 and Day 8 through Day 14
  Blood oxygen level will be measured using the Fitbit Inspire 3 (an actigraphy watch). Sleep Partners of study participants will be asked to wear the actigraphy watch continuously for the 7 days before the participant initiates use of the pillow (Day -7 through Day -1) and continuously for the last 7 days of the participant's pillow use (Day 8 through Day 14).
Change in Partner's physical activity level | Day -7 through Day -1 and Day 8 through Day 14
  Physical activity level will be measured using the Fitbit Inspire 3 (an actigraphy watch). Sleep Partners of study participants will be asked to wear the actigraphy watch continuously for the 7 days before the participant initiates use of the pillow (Day -7 through Day -1) and continuously for the last 7 days of the participant's pillow use (Day 8 through Day 14).
Change in Partner's subjective cognitive function | Baseline and Day 14
  Subjective cognitive function will be measured by a two-question questionnaire: 1) 'How would you rate your memory at the present time? Would you say it is excellent, very good, good, fair, or poor?' and 2) 'Compared to the previous month, would you say your memory is better now, about the same, or worse than it was then?' The two-question questionnaire will be administered prior to the use of the study pillow and again after discontinuing the use of the study pillow.
Change in Partner's objective cognitive function | Baseline and Day 14
  Objective cognitive function will measured by the Montreal Cognitive Assessment (MoCA). The MoCA score ranges from 0-30. A higher score indicates better cognitive function. The MoCA will be administered prior to the use of the study pillow and again after discontinuing the use of the study pillow.

CONTACTS AND LOCATIONS:
Overall Officials: Chang Dae Lee, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rădulescu PV. The Elderly Technically Sleep A Study into the Use of a Smart Breathing Pillow to Improve Sleep in the Elderly Population. 2024;
- [Background] Radwan A, Fess P, James D, Murphy J, Myers J, Rooney M, Taylor J, Torii A. Effect of different mattress designs on promoting sleep quality, pain reduction, and spinal alignment in adults with or without back pain; systematic review of controlled trials. Sleep Health. 2015 Dec;1(4):257-267. doi: 10.1016/j.sleh.2015.08.001. Epub 2015 Oct 19. PMID 29073401
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Ofstedal MB, Fisher GG, Herzog AR. Documentation of Cognitive Functioning Measures in the Health and Retirement Study. 2005. http://hrsonline.isr.umich.edu/sitedocs/userg/dr-006.pdf
- [Background] Chau B. Fitabase makes activity data from Fitbit devices easily accessible for research. iMedicalApps Accessed April 18, 2024. https://www.imedicalapps.com/2016/11/fitbase-fitbit-activity-research/
- [Background] Steffick DE. Documentation of Affective Functioning Measures in the Health and Retirement Study. 2000. http://hrsonline.isr.umich.edu/sitedocs/userg/dr-005.pdf
- [Background] McGuire J. Fitbit Inspire 3 review: the top affordable fitness tracker just got better. Tom's Guide. Accessed April 18, 2024. https://www.tomsguide.com/reviews/fitbit-inspire-3
- [Background] Mollayeva T, Thurairajah P, Burton K, Mollayeva S, Shapiro CM, Colantonio A. The Pittsburgh sleep quality index as a screening tool for sleep dysfunction in clinical and non-clinical samples: A systematic review and meta-analysis. Sleep Med Rev. 2016 Feb;25:52-73. doi: 10.1016/j.smrv.2015.01.009. Epub 2015 Feb 17. PMID 26163057
- [Background] Chung TT, Lee MT, Ku MC, Yang KC, Wei CY. Efficacy of a Smart Antisnore Pillow in Patients with Obstructive Sleep Apnea Syndrome. Behav Neurol. 2021 Jan 14;2021:8824011. doi: 10.1155/2021/8824011. eCollection 2021. PMID 33510821
- [Background] Virk JS, Kotecha B. When continuous positive airway pressure (CPAP) fails. J Thorac Dis. 2016 Oct;8(10):E1112-E1121. doi: 10.21037/jtd.2016.09.67. PMID 27867577
- [Background] Ghadiri M, Grunstein RR. Clinical side effects of continuous positive airway pressure in patients with obstructive sleep apnoea. Respirology. 2020 Jun;25(6):593-602. doi: 10.1111/resp.13808. Epub 2020 Mar 24. PMID 32212210
- [Background] Ramar K, Dort LC, Katz SG, Lettieri CJ, Harrod CG, Thomas SM, Chervin RD. Clinical Practice Guideline for the Treatment of Obstructive Sleep Apnea and Snoring with Oral Appliance Therapy: An Update for 2015. J Clin Sleep Med. 2015 Jul 15;11(7):773-827. doi: 10.5664/jcsm.4858. PMID 26094920
- [Background] Albakri U, Drotos E, Meertens R. Sleep Health Promotion Interventions and Their Effectiveness: An Umbrella Review. Int J Environ Res Public Health. 2021 May 21;18(11):5533. doi: 10.3390/ijerph18115533. PMID 34064108
- [Background] Maness DL, Khan M. Nonpharmacologic Management of Chronic Insomnia. Am Fam Physician. 2015 Dec 15;92(12):1058-64. PMID 26760592
- [Background] Alshaer H, Hummel R, Mendelson M, Marshal T, Bradley TD. Objective Relationship Between Sleep Apnea and Frequency of Snoring Assessed by Machine Learning. J Clin Sleep Med. 2019 Mar 15;15(3):463-470. doi: 10.5664/jcsm.7676. PMID 30853041
- [Background] Senaratna CV, Perret JL, Lodge CJ, Lowe AJ, Campbell BE, Matheson MC, Hamilton GS, Dharmage SC. Prevalence of obstructive sleep apnea in the general population: A systematic review. Sleep Med Rev. 2017 Aug;34:70-81. doi: 10.1016/j.smrv.2016.07.002. Epub 2016 Jul 18. PMID 27568340
- [Background] Elflein J. Share of U.S. adults who snored as of 2022, by age group. Statista. Accessed April 17, 2024.
- [Background] Kara CO, Zencir M, Topuz B, Ardic N, Kocagozoglu B. [The prevalence of snoring in adult population]. Kulak Burun Bogaz Ihtis Derg. 2005;14(1-2):18-24. Turkish. PMID 16227718
- [Background] Garvey JF, Pengo MF, Drakatos P, Kent BD. Epidemiological aspects of obstructive sleep apnea. J Thorac Dis. 2015 May;7(5):920-9. doi: 10.3978/j.issn.2072-1439.2015.04.52. PMID 26101650